CLINICAL TRIAL: NCT05630183
Title: A Randomized, Open-Label, Phase II Trial of Nab-paclitaxel + Gemcitabine With or Without Botensilimab (AGEN1181) in Patients With Metastatic Pancreatic Cancer Who Have Progressed on Prior 5FU + Leucovorin + Irinotecan + Oxaliplatin (FOLFIRINOX)
Brief Title: A Study of Botensilimab in Participants With Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-800-22
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: BOT; 1181; Immunotherapy; Pancreas; Gemcitabine; Nab-paclitaxel
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Combination (Safety Lead-in Phase) (Experimental): Participants will receive botensilimab in combination with standard-of-care chemotherapy (nab-paclitaxel + gemcitabine).
  Interventions: Drug: Botensilimab; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Part 2: Combination (Experimental): Participants will receive botensilimab in combination standard-of-care chemotherapy (nab-paclitaxel + gemcitabine).
  Interventions: Drug: Botensilimab; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Part 2: Standard of Care (Active Comparator): Participants will receive standard-of-care chemotherapy (nab-paclitaxel + gemcitabine).
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Botensilimab — A fully human fragment crystallizable-enhanced monoclonal cytotoxic T lymphocyte antigen 4 antibody administered intravenously.
  Other Names: AGEN1181
  Arms: Part 1: Combination (Safety Lead-in Phase); Part 2: Combination
Drug: Gemcitabine — Standard-of-care chemotherapy administered intravenously.
Drug: Nab-paclitaxel — Standard-of-care chemotherapy administered intravenously.

SUMMARY:
The goal of this clinical trial is to test if the addition of botensilimab to standard chemotherapy improves the efficacy compared to just chemotherapy alone in participants with metastatic pancreatic cancer. One group of participants will only receive chemotherapy while a second group of participants will receive botensilimab and chemotherapy.

DETAILED DESCRIPTION:
This will be a prospective, multicenter, clinical trial of botensilimab in combination with nab-paclitaxel + gemcitabine or nab-paclitaxel + gemcitabine alone. The trial will be conducted in 2 parts. Part 1 will be a safety lead-in to establish the safety and dose of botensilimab for Part 2. Part 2 will be a randomized, open-label assessment of botensilimab (at the dose level determined in Part 1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of pancreatic ductal adenocarcinoma. Note: fine needle aspirate/cytology of tumor in the presence of a pancreatic mass that confirms ductal adenocarcinoma is acceptable.
* Must have had disease progression on any version of FOLFIRINOX for metastatic disease (including onivyde + oxaliplatin + 5-fluorouracil [5-FU] + leucovorin [NALIRIFOX]). Clarification: Participant with initial diagnosis of locally advanced disease may be eligible if upon retrospective review of initial scans, previously unappreciated metastases are able to be identified; Investigator must provide documentation that participant had metastatic disease at the time the participant received FOLFIRINOX. Notes: Progression on a reduced or maintenance fluoropyrimidine based regimen in the metastatic setting is allowed (for example, leucovorin + 5-FU + oxaliplatin [FOLFOX], leucovorin + 5-FU + irinotecan [FOLFIRI], 5-FU, or capecitabine), provided the participant received at least 1 dose of all of the drugs in a FOLFIRINOX regimen.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Life expectancy of at least 3 months.
* Measurable disease on baseline imaging per RECIST 1.1 criteria.
* A < Grade 2 pre-existing peripheral neuropathy per National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0). Because NCI CTCAE v5.0 grading for peripheral neuropathy does not include guidance for "mild" neuropathy, these cases can be graded per the NCI CTCAE v5.0 grading for general adverse events which includes "mild" under Grade 1.
* Acceptable coagulation status as indicated by an international normalized ratio ≤ 1.5 x institutional ULN, except participants on anticoagulation who can be included at the discretion of the investigator.
* Adequate organ function.
* Women of childbearing potential must have a negative urine or serum pregnancy test at screening (within 72 hours of first dose of study drugs).
* Male participants with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study.

Exclusion Criteria:

* Received more than one prior regimen (that is, FOLFIRINOX) for their metastatic disease. (Progression on a reduced or maintenance fluoropyrimidine-based regimen in the metastatic setting is allowed. [for example, FOLFOX, FOLFIRI, 5-FU, or capecitabine], provided the participant received at least 1 dose of all of the drugs in a FOLFIRINOX regimen.)
* History of central nervous system (CNS) metastasis or active CNS metastasis.
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to the first dose of study drugs (that is, participants with a history of prior malignancy are eligible if treatment was completed at least 2 years prior to first dose of study drugs and the participant has no evidence of disease). Participants with history of prior early-stage basal/squamous cell skin cancer or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible.
* Uncontrolled intercurrent illness, including but not limited to clinically significant (that is, active) cardiovascular disease.
* Active, uncontrolled infections, requiring systemic intravenous anti-infective treatment within 2 weeks prior to first dose of study drugs.
* Major surgery within 4 weeks prior to signing of informed consent form (ICF).
* Prior treatment with an immune checkpoint inhibitor.
* Refractory ascites.
* Partial or complete bowel obstruction within the last 3 months prior to signing of ICF, signs/symptoms of bowel obstruction, or known radiologic evidence of impending obstruction.
* Clinically significant gastrointestinal disorders.
* Treatment with one of the following classes of drugs within the delineated time window prior to first dose of study drugs:

  * Cytotoxic agent within 3 weeks or 5 half-lives (whichever is greater).
  * Monoclonal antibodies, antibody-drug conjugates, radioimmunoconjugates, or investigational drug, within 4 weeks, or 5 half-lives, whichever is shorter.
  * Small molecule targeted therapies/tyrosine kinase inhibitors within 14 days or 5 half-lives (whichever is greater).
  * Radiotherapy within 7 days.
* Previous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to first dose of study drugs.
* Received a vaccine, including SARS-CoV-2 vaccine, < 7 days prior to first dose of study drugs.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Symptomatic interstitial lung disease (ILD), history of ILD, or any lung disease which may interfere with detection and management of new immune-mediated pulmonary toxicity.
* History of allogeneic organ transplant.
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 milligrams [mg] daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days prior to the first dose of study drugs. Inhaled or topical steroids, and adrenal replacement steroid doses (≤ 10 mg daily prednisone equivalent), are permitted in the absence of active autoimmune disease.
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years prior to first dose of study drugs (that is, with use of disease-modifying agents or immunosuppressive drugs).
* Pregnant or breastfeeding participants.
* Uncontrolled infection with human immunodeficiency virus.
* Known to be positive for hepatitis B (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection.
* Known active hepatitis C as determined by positive serology and confirmed by polymerase chain reaction.
* Dependence on total parenteral nutrition.
* Participants with concurrent diarrhea > grade 1 at time of randomization despite optimal treatment with standard of care pancreatic enzymes.
* Known active or latent tuberculosis.
* Any condition in the opinion of the principal investigator that might interfere with the participant's participation in the study or in the evaluation of the study results.
* Unwillingness or inability to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival as Assessed by Investigator | Up to 2 years
  Progression-free survival will be defined as the time from the date of randomization to the date of the first objectively documented tumor progression, assessed by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), or death, whichever occurs first.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | First study dose through up 1 year
Overall Survival | Up to 2 years
  Overall survival will be defined as the time from the date of randomization to the date of death due to any cause.
Complete Response | Up to 2 years
  Complete response will be defined by RECIST 1.1 criteria and carbohydrate antigen 19-9 down to normal limits (from at least > 2 x upper limit of normal [ULN]). Cancer antigen 125 or carcinoembryonic antigen will be evaluated for non-expressors of carbohydrate antigen 19-9.
Progression-free Survival as Assessed by Investigator | Up to 2 years
  Progression-free survival will be defined as the time from the date of randomization to the date of the first objectively documented tumor progression, assessed by investigator per RECIST 1.1, or death, whichever occurs first.
Overall Response Rate | Up to 2 years
  Overall response rate will be defined as the proportion of participants whose best overall response is complete response or partial response assessed by investigator per RECIST v1.1.
Duration of Response | Up to 2 years
  Duration of response will be defined as the time from the first determination of an objective response assessed by investigator per RECIST v1.1, until the first documentation of progression or death, whichever occurs first.
Change From Baseline in Carbohydrate Antigen 19-9 | Baseline, 2 years
  Change in carbohydrate antigen 19-9 will be evaluated until progressive disease, death, date of last tumor assessment, or start of new anti-cancer therapy. Cancer antigen 125 or carcinoembryonic antigen will be evaluated for non-expressors of carbohydrate antigen 19-9.
Rates of Normalization of Carbohydrate Antigen 19-9 | Up to 2 years
  Carbohydrate antigen 19-9 normalization will be defined as a value of carbohydrate antigen 19-9 down to normal limits (from at least > 2 x ULN). Cancer antigen 125 or carcinoembryonic antigen will be evaluated for non-expressors of carbohydrate antigen 19-9.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (36):
- United States (36):
  - HonorHealth, Scottsdale, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology, Newport Beach, California
  - UCLA Health - Santa Monica Cancer Care, Santa Monica, California
  - Medical Oncology Hematology Consultants (MOHC) - Helen F. Graham Cancer Center, Newark, Delaware
  - Florida Cancer Specialist South, Fort Myers, Florida
  - Cancer Care Centers of Brevard, Palm Bay, Florida
  - Florida Cancer Specialist North, St. Petersburg, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Maryland Oncology Hematology, Columbia, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Rogel Cancer Center, University of Michigan Medicine, Ann Arbor, Michigan
  - Minnesota Oncology, Minneapolis, Minnesota
  - Nebraska Medicine-Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Summerlin Medical Center II*, Las Vegas, Nevada
  - John Theurer Cancer Center at Hackensack, Hackensack, New Jersey
  - Atlantic Health Systems, Morristown, Morristown, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine Sandra and Edward Meyer Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai Tisch Cancer Institute, New York, New York
  - Oncology Hematology Care - Eastgate, Cincinnati, Ohio
  - Sarah Cannon Research Institute at Tennessee Oncology, Cincinnati, Ohio
  - Lifespan, Providence, Rhode Island
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, Carrollton, Texas
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - TxO - Denison Cancer Center, Denison, Texas
  - The Center for Cancer & Blood Disorders: Fort Worth, Fort Worth, Texas
  - Northeast Texas Cancer & Research Institute, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates - Brock Cancer Center, Norfolk, Virginia
  - Shenandoah Oncology, Winchester, Virginia
  - Swedish Cancer Institute, Seattle, Washington